CLINICAL TRIAL: NCT02303002
Title: Efficacy and Safety of Botulinum Toxin Type A for Injection to Treat Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RT002-CL002; CTA Control No. 179120 (Other: Health Canada); File No. 9427-R1312\1-22C (Other: Health Canada)
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose A (Experimental): Dose A: Botulinum Toxin Type A
  Interventions: Biological: Botulinum Toxin Type A
- Dose B (Experimental): Dose B: Botulinum Toxin Type A
  Interventions: Biological: Botulinum Toxin Type A
- Dose C (Experimental): Dose C: Botulinum Toxin Type A
  Interventions: Biological: Botulinum Toxin Type A
- Dose D (Active Comparator): Dose D: Botulinum Toxin Type A
  Interventions: Biological: Active Comparator botulinum toxin
- Dose E (Placebo Comparator): Dose E: Placebo
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Intramuscular injection (IM)
  Arms: Dose A; Dose B; Dose C
Biological: Active Comparator botulinum toxin — IM injection
  Arms: Dose D
Biological: Placebo Comparator — IM injection
  Arms: Dose E

SUMMARY:
This is a safety and efficacy study of botulinum toxin type A in subjects with glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe glabellar frown lines
* Female or male, 30 to 65 years of age in good general health
* Women of childbearing potential must agree to use an effective method of birth control during the course of the study
* Willing to refrain from receipt of facial fillers, laser treatments or use of products that affect skin remodeling and causes an active dermal response

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to Botulinum Toxin Type A such as amyotrophic lateral sclerosis and motor neuropathy, Lambert-Eaton syndrome, and myasthenia gravis
* Muscle weakness or paralysis, particularly in the treatment area
* Active skin disease or infections or irritation at the treatment area
* Facial asymmetry, deep dermal scarring, or inability to substantially lessen the glabellar frown lines by manually spreading them apart
* Treatment with Botulinum Toxin Type A in the face in the last 6 months or in the last 3 months anywhere in the body

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects assessed as responders by investigator assessment of severity of glabellar lines at maximum frown | Week 24
Duration of response assessed by investigator assessment of severity of glabellar lines at maximum frown from the date of injection to when subject reverts to baseline severity | Up to Week 36

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Bertucci V, Humphrey S, Carruthers J, Solish N, Muhn C, Swift A, Rubio RG, Shears G, Rosen N. Comparing Injectable DaxibotulinumtoxinA and OnabotulinumtoxinA in Moderate and Severe Glabellar Lines: Additional Analyses From a Phase 2, Randomized, Dose-Ranging, Double-Blind, Multicenter Study. Dermatol Surg. 2017 Dec;43 Suppl 3:S262-S273. doi: 10.1097/DSS.0000000000001364. PMID 33065952
- [Derived] Carruthers J, Solish N, Humphrey S, Rosen N, Muhn C, Bertucci V, Swift A, Metelitsa A, Rubio RG, Waugh J, Quiring J, Shears G, Carruthers A. Injectable DaxibotulinumtoxinA for the Treatment of Glabellar Lines: A Phase 2, Randomized, Dose-Ranging, Double-Blind, Multicenter Comparison With OnabotulinumtoxinA and Placebo. Dermatol Surg. 2017 Nov;43(11):1321-1331. doi: 10.1097/DSS.0000000000001206. PMID 28614091